CLINICAL TRIAL: NCT01534598
Title: Phase I Trial of Oral 5-Fluoro-2'-Deoxycytidine With Oral Tetrahydrouridine in Patients With Advanced Solid Tumors
Brief Title: FdCyd and THU for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120066; 12-C-0066
Record Dates: First submitted 2012-02-15; First posted 2012-02-16 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms
Keywords: DNA Methylation; Advanced Cancer; Methyltransferase Inhibitor; Epigenetics; Gene Re-Expression
MeSH Terms: conditions — Neoplasms | interventions — 5-fluoro-2'-deoxycytidine; Tetrahydrouridine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): FdCyd + THU administered on an intermittent schedule in 21-day cycles per dose escalation table. THU will be administered orally at a fixed dose of 3000 mg 30 minutes prior to FdCyd.
  Interventions: Drug: FdCyd + THU

INTERVENTIONS:
Drug: FdCyd + THU — Intravenous FdCyd with THU has been evaluated in a Phase I clinical trial with some preliminary evidence of activity. This trial will investigate oral administration of the drugs, which was shown to be feasible in an expansion cohort of the previous trial.

SUMMARY:
Background:

- FdCyd (also called 5-fluoro-2'-deoxycytidine) and THU (also called tetrahydrouridine) are experimental cancer treatment drugs. FdCyd may change how genes work in cancer cells. THU helps keep FdCyd from being broken down by the body. FdCyd and THU have been given to people on other cancer treatment trials, usually by vein. Researchers want to give FdCyd and THU by mouth to see if they work against cancers that have not responded to earlier treatments.

Objectives:

- To test oral FdCyd and THU on advanced solid tumors that have not responded to earlier treatments.

Eligibility:

- Individuals at least 18 years of age who have advanced solid tumors that have not responded to standard treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies and tumor samples will used to study the cancer before treatment.
* FdCyd and THU will be given in 21-day cycles. THU should be taken 30 minutes before taking FdCyd.
* Participants will take FdCyd and THU by mouth, once a day, for 3 days at the beginning of the first and second weeks of each cycle (days 1 3 and 8 10). The drugs will not be taken during the entire third week of each cycle.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Treatment will continue as long as the cancer is responding to the drugs and serious side effects do not develop.

DETAILED DESCRIPTION:
Background:

* 5-Fluoro-2'-deoxycytidine (FdCyd), a fluoropyrimidine nucleoside analog, has a short (10-minute) half-life and is rapidly degraded in vivo by cytidine deaminase. However, co-administration with tetrahydrouridine (THU), an inhibitor of cytidine/deoxycytidine deaminase, has been shown to increase the AUC of the parent compound more than 4-fold. Increased FdCyd exposure allows it to be taken up intracellularly and converted to its triphosphate, which is incorporated into DNA and inhibits the action of the enzyme DNA methyltransferase (DNMT). Inhibition of DNMT, and in turn DNA methylation, can result in the re-expression of tumor suppressor genes.
* Intravenous FdCyd with THU has been evaluated in a Phase I clinical trial with some preliminary evidence of activity. This trial will investigate oral administration of the drugs, which was shown to be feasible in an expansion cohort of the previous trial.

Primary objectives:

-Establish the safety and tolerability of oral FdCyd in combination with oral THU administered on an intermittent schedule in 21-day cycles to patients with refractory solid tumors

Exploratory objectives:

* Determine the pharmacokinetics of oral FdCyd and oral THU
* Document preliminary evidence of activity of oral FdCyd and oral THU
* Determine the clinical benefit rate (CR+PR+SD at 4 months) in patients treated with study drug combination at the MTD
* Determine effect of study treatment on re-expression of p16 and other select genes silenced by methylation in circulating tumor cells and tumor biopsies
* Evaluate the effect of study treatment on DNA (cytosine-5)-methyltransferase 1 and 3 (DNMT1 and DNMT3) expression in tumor biopsies

Eligibility:

-Adults with histologically documented solid tumors whose disease has progressed after at least one line of standard therapy.

Design:

* This is a multicenter trial with NCI as the coordinating center.
* FdCyd and THU will be administered on an intermittent schedule in 21-day cycles. THU will be administered orally 30 minutes prior to FdCyd.
* The trial will follow a standard Phase I dose escalation design (3-6 patients per cohort).
* Consideration will be given to increasing the days of administration of FdCyd with THU after a target maximum plasma concentration of FdCyd is reached.
* Blood and urine for pharmacokinetic studies will be obtained from all patients. Blood for pharmacodynamic studies will be obtained after we achieve a target Cmax of 1microM.
* Up to 25 patients will be enrolled in the expansion cohort, from which mandatory pre- and post-dose tumor biopsies will be collected for the assessment of pharmacodynamic endpoints, at dose level 8 (160 mg FdCyd + 3000 mg THU 1x daily days 1-6 week 1, days 8-13 week 2, in 21-day cycles).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically documented solid tumors whose disease has progressed on standard therapy that is known to be associated with a survival advantage or have disease for which there is no known standard therapy.
* Patients must have measurable or evaluable disease.
* Diagnosis of malignancy must be confirmed by the department of pathology at the institution where the patient is being enrolled prior to patient enrollment.
* Patients must have completed any chemotherapy, radiation therapy, biologic therapy, or major surgery greater than or equal to 4 weeks prior to enrollment (6 weeks for nitrosoureas or mitomycin C). Patients must be greater than or equal to 2 weeks since any prior administration of a study drug in a Phase 0 or equivalent study, at the discretion of the Principal Investigator. Patients must have recovered to eligibility levels from prior toxicity or adverse events. Patients with bone metastases or hypercalcemia on IV bisphosphonate treatment prior to study entry may continue this treatment.
* Age greater than or equal to18 years. Because no dosing or adverse event data are currently available on the use of FdCyd and THU in patients less than 18 years of age, children are excluded from this study, but may be eligible for future pediatric Phase I combination trials.
* Karnofsky performance status greater than or equal to 60%.
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin less than or equal to 1.5 X institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) greater than or equal to 3 X institutional upper limit of normal
  * creatinine less than 1.5 X institutional upper limit of normal

OR

* creatinine clearance greater than or equal to 60 ML/min for patients with creatinine levels above 1.5 X institutional upper limit of normal

  * Because FdCyd has been shown to be teratogenic in animals, pregnant women are excluded from this trial. Nursing women are also excluded, as there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with FdCyd. Women of childbearing potential must agree to either abstain from sexual intercourse or use two forms of acceptable birth control, including one barrier method, for 4 weeks prior to study entry, for the duration of study participation, and for 3 months after completion of study. Men must use a latex condom every time they have sexual intercourse during therapy and for 3 months after study completion, even if they have had a successful vasectomy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she or her partner should inform the treating physician immediately.
  * Ability to understand and the willingness to sign a written informed consent document.
  * Patients should not be receiving any other investigational agents.
  * Ability to swallow liquids.
  * Willingness to provide blood and urine samples, and biopsy samples if on the expansion phase of the study, for research purposes. For the expansion cohort, patients must have tumor amenable to biospy (excisional or incision biopsies of skin or H & N lesions under visualization) and willingness to undergo a tumor biopsy or patient will be undergoing a procedure due to medical necessity during which the tissue may be collected, or tumor biopsy tissue from a previous research study or medical care is available for submission at registration. Criteria for the submission of tissue are:
* Tissue must have been collected within 3 months prior to registration
* Patient has not received any intervening therapy for their cancer since the collection of the tumor sample
* Tumor tissue must meet the minimum requirements

EXCLUSION CRITERIA:

* Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to active or uncontrolled infection, immune deficiencies, known HIV infection requiring protease inhibitor therapy, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 2 months after treatment of the brain metastases. Patients should be on stable doses of anti-seizure medications. These patients may be enrolled at the discretion of the Principal Investigator.
* History of allergic reactions attributed to fluoropyrimidines (e.g., capecitabine, fluorouracil, fluorodeoxyuridine) or tetrahydrouridine.
* Malabsorption syndrome or other conditions that would interfere with intestinal absorption.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 1 cycle
  FdCyd + THU administered on an intermittent schedule in 21-day cycles per dose escalation table. THU will be administered orally at a fixed dose of 3000 mg 30 minutes prior to FdCyd.

CONTACTS AND LOCATIONS:
Overall Officials: James H Doroshow, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - USC Norris Cancer Center, Los Angeles, California
  - UC Davis Cancer Center, Sacramento, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Penn State, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0066.html